CLINICAL TRIAL: NCT06362668
Title: EU Sites: Fluid Management of Acute Decompensated Heart Failure Subjects Treated With Reprieve Decongestion Management System (DMS) (FASTR-EU)
Brief Title: EU Sites: Fluid Management of Acute Decompensated Heart Failure With Reprieve Decongestion Management System (FASTR-EU)
Acronym: FASTR-EU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reprieve Cardiovascular, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCV-0006-EU
Record Dates: First submitted 2024-02-21; First posted 2024-04-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Diuretics; Furosemide; Bumetanide; Torsemide; Hydrochlorothiazide; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Reprieve Decongestion Management System (Experimental): Subjects randomized to Reprieve System will receive personalized and optimized diuretic and saline infusion using the study device during the course of the treatment.
  Interventions: Device: Reprieve Decongestion Management System
- Optimal Diuretic Therapy (Active Comparator): Sites will consider best practices of optimal diuretic dosing such as those demonstrated in recent randomized trials [Diuretic Strategies in Patients with Acute Heart Failure Trail (DOSE), Acetazolamide in Decompensated Heart Failure with Volume Overload Trial (ADVOR), and Safety and Efficacy of the Combination of Loop with Thiazide-type Diuretics in Patients with Decompensated Heart Failure Trial (CLOROTIC)] for patients randomized to control arm of the trial.
  Interventions: Drug: Diuretic (furosemide, bumetanide, torsemide, hydrochlorothiazide, and/or acetazolamide)

INTERVENTIONS:
Device: Reprieve Decongestion Management System — The Reprieve Decongestion Management System, or Reprieve DMS, is a hospital bedside fluid management console designed to provide personalized and automated infusion of the IV diuretic furosemide and physiological saline in response to the patient's real-time urine output to safely and rapidly decongest patients suffering from Acute Decompensated Heart Failure.
  Arms: Reprieve Decongestion Management System
Drug: Diuretic (furosemide, bumetanide, torsemide, hydrochlorothiazide, and/or acetazolamide) — Best practices of optimal diuretic dosing such as those demonstrated in recent randomized trials (DOSE, ADVOR, CLOROTIC).
  Arms: Optimal Diuretic Therapy

SUMMARY:
The objective of this study is to prospectively compare decongestive therapy administered by the Reprieve DMS system to Optimal Diuretic Therapy (ODT) in the treatment of patients diagnosed with acute decompensated heart failure (ADHF). The main objective is to determine if the Reprieve DMS is non-inferior to state-of-the-art urine sodium guided aggressive diuretic titration in two European HF centers of excellence.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a diagnosis of heart failure as defined by the presence of at least 1 symptom AND 1 sign.
2. ≥10 pounds (4.5 kg) above dry weight either by historical weights or as estimated by health care provider.
3. Prior use of loop diuretics within 30 says prior to admission.
4. ≥ 18 years of age able to provide informed consent and comply with study procedures.

Exclusion Criteria:

1. Inability to place Foley catheter or IV catheter.
2. Hemodynamic instability.
3. Dyspnea due primarily to non-cardiac causes.
4. Acute infection with evidence of systemic involvement.
5. Estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2 calculated using the MDRD equation or current use of renal replacement therapy.
6. Significant left ventricular outflow obstruction, uncorrected complex congenital heart disease, severe stenotic valvular disease, infiltrative or constrictive cardiomyopathy, acute myocarditis, type 1 acute myocardial infarction requiring treatment, or any other pathology that, in the opinion of the investigator, would make aggressive diuresis poorly tolerated.
7. Inability to follow instructions or comply with follow-up procedures.
8. Other concomitant disease or condition that investigator deems unsuitable for the study, including drug or alcohol abuse or psychiatric, behavioral or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the study instructions or follow-up procedures.
9. Severe electrolyte abnormalities.
10. Presence of active coronavirus disease 2019 (COVID-19) infection.
11. Enrollment in another interventional trial during the index hospitalization.
12. Inability to return for follow-up study visits.
13. Life expectancy less than 3 months.
14. Women who are pregnant or intend to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Total sodium loss (in mmol of sodium) per 24 hours | End of treatment, an average of 72 hours
  Primary efficacy endpoint is total sodium loss in mmol of sodium at end of randomized therapy normalized to 24 hours (up to a maximum of 72 hours).
Comparison of occurrence of composite endpoint comprised of clinically significant acute kidney injury, severe electrolyte abnormality, or symptomatic hypotension or hypertensive emergency. | Through study completion, an average of 90 days
  Primary safety endpoint is positive if any of the following occurs in an individual participant:
  1. Clinically significant acute kidney injury defined as Kidney Disease-Improving Global Outcomes (KDIGO) stage 2 or greater Acute Kidney Injury (AKI) [≥ doubling of baseline serum creatinine or use of renal replacement therapy (RRT)]
  2. Severe electrolyte abnormality defined as serum potassium <3.0 milliequivalent/liter (mEq/L), magnesium <1.3 mEq/L, or sodium <135 mEq
  3. Symptomatic hypotension (systolic pressure <80mmHg) or hypertensive (systolic pressure >200 mmHg and/or diastolic pressure >120 mmHg) emergency.

SECONDARY OUTCOMES:
Total net fluid volume loss (difference between urine output volume and fluid input volume) per 24 hours | End of treatment, an average of 72 hours
  Difference between volume of urine output and fluid input during primary treatment normalized to 24 hours.
Weight loss per 24 hours at end of randomized therapy | End of treatment, an average of 72 hours
  Total time on loop diuretics during primary treatment
Time on IV loop diuretic | End of treatment, an average of 72 hours
  Total time on loop diuretics from initiation of randomized therapy to last dose of IV loop diuretic administered for ADHF
Number of participants with ≥ 0.3 mg/dL increase in serum creatinine | End of treatment, an average of 72 hours
  In hospital worsening renal function defined as ≥ 0.3 mg/dL increase in serum creatinine during randomized therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- University Medical Center Groningen, Groningen, Netherlands
- Wroclaw Medical University, Wroclaw, Poland

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT06362668/SAP_000.pdf